CLINICAL TRIAL: NCT03826550
Title: A Randomized, Double-Blind, Placebo-Controlled, Three-Arm, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Diclofenac Sodium Gel 3% (Encube Ethicals) Compared to Solaraze® (Diclofenac Sodium) Gel 3% (Fougera Pharmaceuticals Inc.) in the Treatment of Actinic Keratosis
Brief Title: Therapeutic Equivalence of Diclofenac Sodium Gel 3% vs Solaraze ® in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Encube Ethicals Pvt. Ltd. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENC16102
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Diclofenac; Gels

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, three-arm, parallel group, multiple-site bioequivalence study with clinical endpoints.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study products are blinded and provided to the patients in the same packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diclofenac Sodium Gel3% (Experimental): Diclofenac Sodium Gel 3%, dosed twice daily for 60 days.
  Interventions: Drug: Diclofenac Sodium Gel
- Solaraze (Active Comparator): Solaraze Gel dosed twice daily for 60 days.
  Interventions: Drug: Solaraze 3% Topical Gel
- Placebo (Placebo Comparator): Placebo Gel dosed twice daily for 60 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diclofenac Sodium Gel — Twice daily for 60 days. Each patient is expected to receive 120 doses
  Arms: Diclofenac Sodium Gel3%
Drug: Solaraze 3% Topical Gel — Twice daily for 60 days. Each patient is expected to receive 120 doses
  Arms: Solaraze
Other: Placebo — Twice daily for 60 days. Each patient is expected to receive 120 doses
  Arms: Placebo

SUMMARY:
Therapeutic Equivalence of Diclofenac Sodium Gel 3% and Solaraze ®, in the treatment of Actinic Keratosis

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Three-Arm, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Diclofenac Sodium Gel 3% (Encube Ethicals) Compared to Solaraze® (diclofenac sodium) Gel 3% (Fougera Pharmaceuticals Inc.) in the Treatment of Actinic Keratosis

ELIGIBILITY:
Inclusion Criteria:

1. Signed Institutional Review Board (IRB)-approved informed consent form that meets all criteria of current Food and Drug Administration regulations.
2. Male or non-pregnant, non-lactating female, 18 years of age or older.
3. Diagnosis of AK with at least five and no more than ten clinically typical, visible, discrete, non-hyperkeratotic, non-hypertrophic AK lesions, each at least 4 mm in diameter, contained within a contiguous 25 cm2 treatment area on the face and/or bald scalp.
4. Females of childbearing potential must not be pregnant or lactating at Visit 1 (as confirmed by a negative urine pregnancy test with a sensitivity of less than 50 mIU/ mL or equivalent units of human chorionic gonadotropin). Women of childbearing potential must agree to the use of a reliable method of contraception (e.g., total abstinence, intrauterine device, a double-barrier method, oral, transdermal, injected, or implanted non-hormonal or hormonal contraceptive) throughout the study. Female patients using hormonal contraceptives should have been on the same product/dosing regimen for at least 28 days before Visit 1 and should not change this regimen during the study. A sterile sexual partner is not considered an adequate form of birth control.
5. Skin pigmentation that will allow discernment of erythema.

Exclusion Criteria:

1. Females who are pregnant, lactating or planning to become pregnant during the study period.
2. Active gastrointestinal ulceration or bleeding.
3. Current evidence or history of severe renal or hepatic impairment.
4. Known allergy or hypersensitivity to diclofenac, benzyl alcohol, polyethylene glycol monomethyl ether 359, hyaluronate sodium or other excipients in the test, reference or vehicle gel.
5. Known allergy or hypersensitivity to other NSAIDs, including aspirin.
6. Presence of atopic dermatitis, basal cell carcinoma, squamous cell carcinoma, eczema, psoriasis, rosacea, sunburn, exfoliative dermatitis, open or recent skin wounds, active infections or other possible skin conditions on the face or bald scalp that in the Investigator's opinion would interfere with the study assessments or put the patient at risk.
7. Use of oral isotretinoin within six months before randomization.
8. Use within six months before Visit 1 on the face or bald scalp of 1) chemical peel, 2) dermabrasion, 3) laser abrasion, 4) PUVA (psoralen plus ultraviolet A) therapy, or 5) UVB therapy.
9. Use within one month before Visit 1 on the face or bald scalp of 1) cryodestruction or chemodestruction, 2) curettage, 3) photodynamic therapy, 4) surgical excision, 5) topical 5-fluorouracil, 6) topical corticosteroids, 7) topical diclofenac, 8) topical imiquimod, 9) topical retinoids, or 10) other treatments for AK including glycolic acids or over the- counter (OTC) products containing retinol, alpha or beta hydroxy acids. The occasional use of ophthalmic, intranasal or inhaled corticosteroids (e.g., management of allergic conjunctivitis) is acceptable and not reason for exclusion. Use of inhaled corticosteroids for the management of chronic and stable conditions (e.g., persistent asthma and chronic obstructive pulmonary disease [COPD]) is acceptable as long as it has been on a stable dose for a minimum of three months before the start of the study and up to 1 mg/day.
10. Use within one month before Visit 1 of 1) immunomodulators or immunosuppressive therapies, 2) interferon, 3) systemic corticosteroids or 4) cytotoxic drugs.
11. Receipt of 5-Fluorouracil or other systemic cancer chemotherapy within 6 months before Visit 1.
12. Any condition, medical, psychological, or social, that, in the Investigator's opinion, would interfere with participation in the study or put the patient at risk.
13. Inability to understand the requirements of the study and the relative information or are unable or not willing to comply with the study protocol.
14. Receipt of any drug as part of a research study within 30 days before Visit 1.
15. Employees of the Investigator or research center or their immediate family members.
16. Patients who have participated in this study previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
proportion of patients in each treatment group with 100% clearance of all AK Lesions | Day 90 (30 days after completion of a 60 day treatment)
Superiority of the test and reference products against the placebo | Day 90 (30 days after completion of a 60 day treatment)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Dermatology Trial Associates, Bryant, Arkansas
  - West Coast Research, San Ramon, California
  - Universal Medical and Research Center, LLC, Coral Gables, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Multi-Speciality Research Associates, Inc., Lake City, Florida
  - FXM Research, Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Moore Clinical Research, Tampa, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - DS Research, New Albany, Indiana
  - DS Research, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - DTRL, Inc., Henderson, Nevada
  - Dermatology Consulting Services, High Point, North Carolina
  - Sterling Research Group, Cincinnati, Ohio
  - DermDox Centers for Dermatology, Hazleton, Pennsylvania
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
  - Anderson Dermatology, Anderson, South Carolina
  - Greenville Dermatology, LLC, Greenville, South Carolina
  - Sirius Clinical Research, LLC, Austin, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No